CLINICAL TRIAL: NCT05175248
Title: A Randomized Controlled Trial of a Nutritional Intervention for Endometriosis
Brief Title: Nutritional Intervention for Endometriosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00059650
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
Keywords: endometriosis; plant-based; vegan; low-fat; diet; nutrition
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-based Intervention Group (Experimental): Intervention group participants will adopt a low-fat, plant-based diet for 12 weeks. Participants will be provided with a commercially available supplement containing 100 micrograms of vitamin B12 and asked to take it daily during the study. Alcoholic beverages will be limited to 1 per day. Participants will be asked to keep their physical activity level constant.
  Interventions: Behavioral: Plant-based Intervention Group
- Control Group (No Intervention): Control group participants will be asked to maintain their usual diet for the duration of the 12-week study period. Participants will be provided with a commercially available supplement containing 100 micrograms of vitamin B12 and asked to take it daily during the study. Alcoholic beverages will be limited to 1 per day. Participants will be asked to keep their physical activity level constant. At the conclusion of the 12 weeks, control group participants will be offered instruction in the plant-based diet.

INTERVENTIONS:
Behavioral: Plant-based Intervention Group — Participants in the intervention group will be instructed in ways to adopt a plant-based diet, use appropriate methods of food preparation, and make meals enjoyable and appetizing. The plant-based diet primarily emphasizes whole grains, vegetables, beans and legumes, and fruits. Animal products and added oils will be proscribed and the use of ultra-processed foods, sugar, and sugar-sweetened beverages will be discouraged. Fat intake will be limited to 20-30 g/day.
  Arms: Plant-based Intervention Group

SUMMARY:
In a 12-week parallel study, women with a verified diagnosis of endometriosis will be randomly assigned to follow a low-fat plant-based diet or to stay on their usual diets for 12 weeks. Participants in both groups will be asked to make no changes to their exercise patterns for the study period. Changes in pain, quality of life, and inflammatory biomarkers from baseline to final will be the primary outcomes. Secondary outcomes will include changes in body weight, blood lipids, gut microbiome composition, and hormonal changes.

DETAILED DESCRIPTION:
Endometriosis is a chronic, painful condition that affects 5-10% of reproductive aged women. It is characterized by the presence of endometrial cells outside the uterus, causing pain and infertility. Current therapies to temporarily control symptoms include surgery and medical options with significant side effects. Women with endometriosis may have several surgeries by their mid-20s. The medical costs associated with endometriosis in the US alone are about $3.6 billion annually, and the total annual health care cost associated with endometriosis in 2002 was $22 billion, one-third of which is direct health care costs, with two-thirds attributed to loss of productivity.

Diet may play important roles in endometriosis through its effect on circulating estrogen concentrations and inflammatory processes. Reduced fat intake and increased fiber intake have been shown to reduce estrogen levels, a key determinant of endometriosis activity. Some evidence suggests a pathogenic role for the gut microbiome, which influences the mucosal immune system and pelvic inflammation. The microbiome is responsive to short term dietary intervention, although long term changes have not been well characterized.

Therefore, the investigators propose a novel intervention strategy using a plant-based diet to improve pain, inflammation, and quality of life.

The morbidity caused by endometriosis is substantial in terms of pain, reduced quality of life, lost productivity, and effects on relationships. Current medical therapies are limited in efficacy and have major side effects. Typical palliative surgery does not cure endometriosis. Better understanding of diet's ability to influence the disease process has the potential to improve quality of life and daily functioning without the cost and side effects of current therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a surgical, imaging, or clinical diagnosis of endometriosis
2. Age 18-45 years
3. Stable health condition and medications for past 3 months
4. Modified Biberoglu and Behrman (B&B) pelvic pain score of at least 5/9
5. Able to follow a plant-based diet for 12 weeks
6. Willing to be randomly assigned to either a plant-based group or a control group that will not make any dietary changes for 12 weeks

Exclusion Criteria:

1. Body mass index ≥ 40 kg/m2
2. Smoking or drug abuse during the past six months
3. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
4. Unstable medical or psychiatric illness
5. Already following a plant-based diet
6. Pregnant or breastfeeding, or plans of pregnancy within the study period
7. Hysterectomy or ovariectomy
8. Fibroids, ovarian cysts, pelvic inflammatory disease
9. Endocrine inflammatory conditions, such as Cushing's syndrome, Hashimoto's thyroiditis, Graves' disease, type 1 diabetes mellitus, and Addison's disease
10. Lack of English fluency
11. Unable or unwilling to participate in all components of the study
12. Evidence of an eating disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Modified Biberoglu and Behrman Scale: change from baseline | at baseline and at 12 weeks
  Endometriosis-specific pain scale will be used. For inclusion in study, participants require a score of at least 5/9.
Endometriosis Health Profile (EHP-30): change from baseline | at baseline and at 12 weeks
  The EHP-30 questionnaire is the only validated quality of life questionnaire for the use in endometriosis.
Inflammatory biomarkers: change from baseline | at baseline and at 12 weeks
  Blood tests for biomarkers of inflammation (hsCRP, TNF-alpha, IL-1 beta and IL-6).

SECONDARY OUTCOMES:
Body weight: change from baseline | at baseline and at 12 weeks
  Weight will be measured using a self-calibrating scale (Renpho).
Blood lipids: change from baseline | at baseline and at 12 weeks
  Change in blood lipids assessed via blood tests including lipid panels.
Estrogen levels: change from baseline | at baseline and at 12 weeks
  Estradiol, free estradiol, and sex hormone binding globulin (SHBG) will be measured through blood tests.
Gut microbiome composition: change from baseline | at baseline and at 12 weeks
  Participants will collect stool samples for microbiome analysis. Sample collection will be carried out using home collection procedures with samples returned through local post. The participants will apply a small smear to the tips of a swab from used toilet paper. The swab will, in turn, be used to transfer the smear to a fecal occult blood test (FOBT) card that will be returned by mail to a laboratory for analysis.
Biomarkers of endometriosis and inflammation: change from baseline | at baseline and at 12 weeks
  Plasma levels of brain-derived neurotrophic factor (BDNF) and IL-10 will be measured through blood tests.

CONTACTS AND LOCATIONS:
Overall Officials: Hana Kahleova, MD, PhD, Principal Investigator — Physicians Committee for Responsible Medicine; Neal Barnard, MD, Study Director — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Kennedy S, Bergqvist A, Chapron C, D'Hooghe T, Dunselman G, Greb R, Hummelshoj L, Prentice A, Saridogan E; ESHRE Special Interest Group for Endometriosis and Endometrium Guideline Development Group. ESHRE guideline for the diagnosis and treatment of endometriosis. Hum Reprod. 2005 Oct;20(10):2698-704. doi: 10.1093/humrep/dei135. Epub 2005 Jun 24. PMID 15980014
- [Background] Khanaki K, Nouri M, Ardekani AM, Ghassemzadeh A, Shahnazi V, Sadeghi MR, Darabi M, Mehdizadeh A, Dolatkhah H, Saremi A, Imani AR, Rahimipour A. Evaluation of the relationship between endometriosis and omega-3 and omega-6 polyunsaturated fatty acids. Iran Biomed J. 2012;16(1):38-43. doi: 10.6091/ibj.1025.2012. PMID 22562031
- [Background] Marik JJ. Leuprolide acetate depot and hormonal add-back in endometriosis: a 12-month study. Obstet Gynecol. 1998 May;91(5 Pt 1):793-4. doi: 10.1097/00006250-199805000-00029. No abstract available. PMID 9572232
- [Background] Stratton P, Sinaii N, Segars J, Koziol D, Wesley R, Zimmer C, Winkel C, Nieman LK. Return of chronic pelvic pain from endometriosis after raloxifene treatment: a randomized controlled trial. Obstet Gynecol. 2008 Jan;111(1):88-96. doi: 10.1097/01.AOG.0000297307.35024.b5. PMID 18165396
- [Background] Rogers PA, D'Hooghe TM, Fazleabas A, Giudice LC, Montgomery GW, Petraglia F, Taylor RN. Defining future directions for endometriosis research: workshop report from the 2011 World Congress of Endometriosis In Montpellier, France. Reprod Sci. 2013 May;20(5):483-99. doi: 10.1177/1933719113477495. Epub 2013 Feb 20. PMID 23427182
- [Background] Goldin BR, Woods MN, Spiegelman DL, Longcope C, Morrill-LaBrode A, Dwyer JT, Gualtieri LJ, Hertzmark E, Gorbach SL. The effect of dietary fat and fiber on serum estrogen concentrations in premenopausal women under controlled dietary conditions. Cancer. 1994 Aug 1;74(3 Suppl):1125-31. doi: 10.1002/1097-0142(19940801)74:3+3.0.co;2-5. PMID 8039147
- [Background] Sender R, Fuchs S, Milo R. Revised Estimates for the Number of Human and Bacteria Cells in the Body. PLoS Biol. 2016 Aug 19;14(8):e1002533. doi: 10.1371/journal.pbio.1002533. eCollection 2016 Aug. PMID 27541692
- [Background] Gill SR, Pop M, Deboy RT, Eckburg PB, Turnbaugh PJ, Samuel BS, Gordon JI, Relman DA, Fraser-Liggett CM, Nelson KE. Metagenomic analysis of the human distal gut microbiome. Science. 2006 Jun 2;312(5778):1355-9. doi: 10.1126/science.1124234. PMID 16741115
- [Background] Longman RS, Littman DR. The functional impact of the intestinal microbiome on mucosal immunity and systemic autoimmunity. Curr Opin Rheumatol. 2015 Jul;27(4):381-7. doi: 10.1097/BOR.0000000000000190. PMID 26002030
- [Background] Hooper LV, Littman DR, Macpherson AJ. Interactions between the microbiota and the immune system. Science. 2012 Jun 8;336(6086):1268-73. doi: 10.1126/science.1223490. Epub 2012 Jun 6. PMID 22674334
- [Background] Ivanov II, Frutos Rde L, Manel N, Yoshinaga K, Rifkin DB, Sartor RB, Finlay BB, Littman DR. Specific microbiota direct the differentiation of IL-17-producing T-helper cells in the mucosa of the small intestine. Cell Host Microbe. 2008 Oct 16;4(4):337-49. doi: 10.1016/j.chom.2008.09.009. PMID 18854238
- [Background] Wu HJ, Ivanov II, Darce J, Hattori K, Shima T, Umesaki Y, Littman DR, Benoist C, Mathis D. Gut-residing segmented filamentous bacteria drive autoimmune arthritis via T helper 17 cells. Immunity. 2010 Jun 25;32(6):815-27. doi: 10.1016/j.immuni.2010.06.001. PMID 20620945
- [Background] Mazmanian SK, Liu CH, Tzianabos AO, Kasper DL. An immunomodulatory molecule of symbiotic bacteria directs maturation of the host immune system. Cell. 2005 Jul 15;122(1):107-18. doi: 10.1016/j.cell.2005.05.007. PMID 16009137
- [Background] Mazmanian SK, Round JL, Kasper DL. A microbial symbiosis factor prevents intestinal inflammatory disease. Nature. 2008 May 29;453(7195):620-5. doi: 10.1038/nature07008. PMID 18509436
- [Background] Fredricks DN, Fiedler TL, Marrazzo JM. Molecular identification of bacteria associated with bacterial vaginosis. N Engl J Med. 2005 Nov 3;353(18):1899-911. doi: 10.1056/NEJMoa043802. PMID 16267321
- [Background] Ravel J, Gajer P, Abdo Z, Schneider GM, Koenig SS, McCulle SL, Karlebach S, Gorle R, Russell J, Tacket CO, Brotman RM, Davis CC, Ault K, Peralta L, Forney LJ. Vaginal microbiome of reproductive-age women. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4680-7. doi: 10.1073/pnas.1002611107. Epub 2010 Jun 3. PMID 20534435
- [Background] Srinivasan S, Hoffman NG, Morgan MT, Matsen FA, Fiedler TL, Hall RW, Ross FJ, McCoy CO, Bumgarner R, Marrazzo JM, Fredricks DN. Bacterial communities in women with bacterial vaginosis: high resolution phylogenetic analyses reveal relationships of microbiota to clinical criteria. PLoS One. 2012;7(6):e37818. doi: 10.1371/journal.pone.0037818. Epub 2012 Jun 18. PMID 22719852
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Agarwal SK, Chapron C, Giudice LC, Laufer MR, Leyland N, Missmer SA, Singh SS, Taylor HS. Clinical diagnosis of endometriosis: a call to action. Am J Obstet Gynecol. 2019 Apr;220(4):354.e1-354.e12. doi: 10.1016/j.ajog.2018.12.039. Epub 2019 Jan 6. PMID 30625295
- [Background] Practice bulletin no. 114: management of endometriosis. Obstet Gynecol. 2010 Jul;116(1):223-236. doi: 10.1097/AOG.0b013e3181e8b073. No abstract available. PMID 20567196
- [Background] Ridout MS. Testing for random dropouts in repeated measurement data. Biometrics. 1991 Dec;47(4):1617-9; discussion 1619-21. PMID 1786335
- [Background] Paik, MC, Quasi-likelihood regression models with missing covariates, Biometrika 1996: Vol. 83, No. 4., 825-834
- [Background] Gibbons RD, Hedeker D, Waternaux C, Davis JM. Random regression models: a comprehensive approach to the analysis of longitudinal psychiatric data. Psychopharmacol Bull. 1988;24(3):438-43. No abstract available. PMID 3153505
- [Background] Hedeker D, Gibbons R, Waternaux C. Sample size estimation for longitudinal designs with attrition: Comparing time-related contrasts between two groups. Journal of Educational and Behavioral Statistics. 1999; 24:70-93.
- [Background] Westfall PH and Young SS. (1993). Resampling-based Multiple Testing: Examples and Methods for Multiple P-value Adjustment. John Wiley & Sons: New York.